CLINICAL TRIAL: NCT03284892
Title: Screen and Intervene: A Diagnostic Accuracy Study and A Randomized, Open-label, Controlled Trial for Postextubation Dysphagia
Brief Title: Screening and Intervention of Postextubation Dysphagia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Taiwan University Hospital (Other)
Collaborators: Ministry of Science and Technology, Taiwan (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 201705051RIND
Record Dates: First submitted 2017-08-21; First posted 2017-09-15 (Actual); Last update posted 2023-07-20 (Actual); Status verified 2020-08

CONDITIONS: Oropharyngeal Dysphagia; Swallowing Disorder; Randomized Controlled Trial; Endotracheal Intubation
Keywords: postextubation dysphagia; endotracheal intubation; randomized controlled trial; dysphagia intervention; dysphagia screening
MeSH Terms: conditions — Deglutition Disorders

STUDY DESIGN:
Intervention Model Description: Qualified participants will receive a two-item screening and FEES examination within 48 hours postextubation. Then participants will be randomly assigned, on a 1:1 ratio, to an intervention, SOC group or a control group (receiving usual care). A research nurse will provide the SOC program for seven days or until death or hospital discharge. All outcomes, including resumption of oral feeding, incidence of pneumonia, and incidence of penetration and aspiration, will be evaluated by an independent outcome assessor.
Who Masked: Care Provider, Investigator, Outcomes Assessor
Masking Description: To maintain allocation concealment, the investigators ensured that only the intervention nurse had access to the random sequence. Physicians and staff at the study sites were aware of a pending nursing-intervention study but were blinded with respect to the hypothesis, group allocation, specific SOC protocols, and study endpoints. Moreover, outcome assessors were blinded to the group assignments, ensuring an unbiased evaluation.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- SOC group (Experimental): Received SOC program addition to usual care
  Interventions: Behavioral: SOC program
- Control group (No Intervention): Received usual care only

INTERVENTIONS:
Behavioral: SOC program — A once-daily, 7-day SOC program, including oral-motor exercise, sensory stimulation and lubrication, and safe-swallowing education.
  Arms: SOC group

SUMMARY:
This clinical trial aims to test the validity of a two-item swallowing screen and to examine the effects of the Swallowing and Oral-Care (SOC) Program on resumption of oral intake, incidence of penetration and aspiration, and incidence of pneumonia in adult patients who successfully extubated after ≥ 48 hours of endotracheal intubation.

DETAILED DESCRIPTION:
Endotracheal intubation is life-sustaining, but it may contribute to postextubation dysphagia (PED) increasing the risk of penetration, aspiration, and aspiration pneumonia. Up to 84% of extubated patients had PED and approximately 60% penetrated and aspirated that can lead to aspiration pneumonia. The aims of this three-year, two-stage study are: 1) In the first stage, the investigators develop a two-item swallowing screen involving oral stereognosis and cough reflex test for predicting the resumption of oral intake and feeding-tube dependence by using a diagnostic accuracy study method; 2) In the second stage, the investigators conduct a randomized, open-label, controlled trial design to examine the effect of a once-daily, 7-day SOC Program on resumption of oral intake, incidence of penetration and aspiration, and incidence of pneumonia in adult patients who successfully extubated after ≥ 48 hours of endotracheal intubation.

ELIGIBILITY:
Inclusion Criteria:

* Patient who is over 20 years old.
* Patient how has received over 48 hours endotracheal intubation and had been successfully extubated.

Exclusion Criteria:

* Patient who has a history of neuromuscular disease (e.g., parkinsonism or stroke) or head and neck deformities.
* Patient who has preexisting difficulty swallowing.
* Patient who has received a tracheostomy.
* Patient who were unable to follow verbal instructions.
* Patient who were on contact and droplet precautions (e.g., open tuberculosis)
* Patient who were receiving continuous noninvasive ventilation after extubation that precluded the delivery of an SOC intervention

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 145 (Actual)
Dates: Start 2017-09-19 (Actual); Primary Completion 2020-08-08 (Actual); Study Completion 2020-08-08 (Actual)

PRIMARY OUTCOMES:
Resumption of oral feeding | Postextubation 7 days
  Measured by Functional Oral Intake Scale
Incidence of penetration and aspiration | Time points of assessments: within 48 hrs postextubation and at the day 10 postextubation
  Measured by the Fiberoptic endoscopic evaluation of swallowing (FEES) with optional and the study participants either opt-in or opt-out for this procedure, given that its invasive-nature procedure.
Incidence of pneumonia | Postextubation 30 days
  Abstracted from electronic medical records, based on the American Thoracic Society/Infectious Diseases Society of America criteria.

SECONDARY OUTCOMES:
Incidence of feeding tube dependency | Postextubation 30 days
  Abstracted from electronic medical records
Unstimulated salivary flow rate (centimeter/5 minutes) | Time points of assessments: within 48 hours postextubation and at the day 10 postextubation
  Measured by the whatman 41 test strip
Oral health status score | Time points of assessments: within 48 hours postextubation and at the day 10 postextubation
  Measured by the oral Assessment Guide
Lip closure and lingual diadochokinetic status | Time points of assessments: within 48 hours postextubation and at the day 10 postextubation
  Measured by the Frenchay Dysarthria Assessment

CONTACTS AND LOCATIONS:
Overall Officials: Cheryl Chia-Hui Chen, Prof., Principal Investigator — School of Nursing, College of Medicine, National Taiwan University
Locations (1):
- National Taiwan University Hospital, Taipei, Taiwan

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Siao SF, Ku SC, Tseng WH, Wei YC, Chang YC, Hsiao TY, Wang TG, Chen CC. Effects of a swallowing and oral-care program on resuming oral feeding and reducing pneumonia in patients following endotracheal extubation: a randomized, open-label, controlled trial. Crit Care. 2023 Jul 12;27(1):283. doi: 10.1186/s13054-023-04568-6. PMID 37438759
- [Derived] Siao SF, Tseng WH, Wang TG, Wei YC, Hsiao TY, Ku SC, Chen CC. Predicting feeding-tube dependence in patients following endotracheal extubation: a two-item swallowing screen. BMC Pulm Med. 2021 Dec 6;21(1):403. doi: 10.1186/s12890-021-01771-5. PMID 34872549